CLINICAL TRIAL: NCT04221477
Title: A Phase III, Randomized, Double-Blind, Placebo-Controlled, Multicenter Study to Evaluate the Efficacy and Safety of Obinutuzumab in Patients With ISN/RPS 2003 Class III or IV Lupus Nephritis
Brief Title: A Study to Evaluate the Efficacy and Safety of Obinutuzumab in Participants With ISN/RPS 2003 Class III or IV Lupus Nephritis
Acronym: REGENCY
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CA41705; 2019-004034-42 (EudraCT Number); 2023-503628-22-00 (EU CTIS Number)
Record Dates: First submitted 2020-01-07; First posted 2020-01-09 (Actual); Results first posted 2025-11-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Lupus Nephritis
MeSH Terms: conditions — Lupus Nephritis | interventions — obinutuzumab; Prednisone; Methylprednisolone; Acetaminophen; Diphenhydramine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Obinutuzumab (Experimental): Participants will be randomized into 2 groups. Group 1 will receive obinutuzumab 1000 mg IV at baseline and Weeks 2, 24, 26, 50, and 52 plus MMF and oral prednisone. Group 2 receive obinutuzumab 1000 mg IV at baseline and Weeks 2, 24, 26, and 52 plus MMF and oral prednisone. Group 2 participants will receive a placebo infusion at their Week 50 visit.
  Participants with an adequate response at Week 76 will continue receiving blinded obinutuzumab infusions every 6 months starting at Week 80.
  Participants without an adequate response at Week 76 may be eligible for open-label obinutuzumab starting at Week 80.
  After study unblinding, participants may be eligible for further open-label obinutuzumab treatment.
  Interventions: Drug: Obinutuzumab; Drug: MMF; Drug: Prednisone; Drug: Methylprednisolone; Drug: Acetaminophen; Drug: Diphenhydramine
- Placebo (Placebo Comparator): Placebo participants will receive obinutuzumab matched placebo at baseline and Weeks 2, 24, 26, 50, and 52 plus MMF and oral prednisone.
  Participants with an adequate response at Week 76 will continue receiving blinded obinutuzumab infusions every 6 months starting at Week 80.
  Participants without an adequate response at Week 76 may be eligible for open-label obinutuzumab starting at Week 80.
  After study unblinding, participants may be eligible for further open-label obinutuzumab treatment.
  Interventions: Drug: Obinutuzumab; Drug: MMF; Drug: Prednisone; Drug: Placebo; Drug: Methylprednisolone; Drug: Acetaminophen; Drug: Diphenhydramine

INTERVENTIONS:
Drug: Obinutuzumab — Obinutuzumab will be administered by IV infusion at a dose of 1000 mg at Baseline and Weeks 2, 24, 26, 50 (group 2: placebo), and 52 and subsequently from Week 80 and every 6 months thereafter, based on response.
  Other Names: Gazyva, GA101, RO5072759
Drug: MMF — MMF willl be administered at a target dose of 2.0 - 2.5 g/day in divided doses through Week 80.
Drug: Prednisone — Prednisone 0.5 mg/kg/day (maximum 60 mg/day) will be started on Day 2. Beginning on Day 15, prednisone will be tapered to 5 mg/day and continued until Week 80.
Drug: Placebo — Placebo matching obinutuzumab will be administered by IV infusion at baseline and Weeks 0, 2, 24, 26, 50 and 52 and subsequently from Week 80 and every 6 months thereafter based on response.
  Arms: Placebo
Drug: Methylprednisolone — Methylprednisolone 80 mg IV will be administered as predmedication prior to infusions.
Drug: Acetaminophen — Acetaminophen 650-1000 mg will be administered as premedication prior to infusions.
Drug: Diphenhydramine — Diphenhydramine 50 mg will be administered as premedication prior to infusions.

SUMMARY:
This study will evaluate the efficacy, safety, and pharmacokinetics of obinutuzumab compared with placebo in participants with International Society of Nephrology/Renal Pathology Society (ISN/RPS) 2003 class III or IV lupus nephritis (LN) when added on to standard-of-care therapy consisting of mycophenolate mofetil (MMF) and corticosteroids.

ELIGIBILITY:
Key Inclusion Criteria:

* Diagnosis of active or active/chronic ISN/RPS 2003 Class III or IV proliferative LN as evidenced by renal biopsy performed within 6 months. Participants may co-exhibit Class V disease in addition to either Class III or Class IV disease
* Urine protein to creatinine ratio greater than or equal to (>/=) 1 on a 24-hour collection
* Other inclusion criteria may apply

Key Exclusion Criteria:

* Pregnancy or breastfeeding
* Severe renal impairment or the need for dialysis or renal transplantation
* Receipt of an excluded therapy, including any anti-CD20 therapy less than 9 months prior to screening or during screening; or cyclophosphamide, tacrolimus, ciclosporin, or voclosporin during the 2 months prior to screening or during screening
* Significant or uncontrolled medical disease which, in the investigator's opinion, would preclude participant participation
* Known active infection of any kind or recent major episode of infection
* Intolerance or contraindication to study therapies
* Other exclusion criteria may apply

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 271 (Actual)
Dates: Start 2020-08-10 (Actual); Primary Completion 2024-08-15 (Actual); Study Completion 2031-02-28 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (74):
- United States (18):
  - University of Alabama at Birmingham Medical Center, Birmingham, Alabama
  - Wallace Rheumatic Study Center, Beverly Hills, California
  - Kaiser Permanente - Fontana, Fontana, California
  - Kaiser Permanente - San Francisco Medical Center, San Francisco, California
  - Stanford University Medical Center, Stanford, California
  - Univ Colorado Health Sci Ctr, Aurora, Colorado
  - Yale Medical Group, New Haven, Connecticut
  - University of Miami Miller School of Medicine, Miami, Florida
  - Georgia Nephrology, Lawrenceville, Georgia
  - North Shore University Hospital, Manhasset, New York
  - NYU Langone Medical Center, New York, New York
  - Columbia University Medical Center, New York, New York
  - AD-CARE, University of Rochester Medical Center, Rochester, New York
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - Oklahoma Medical Research Foundation, Oklahoma City, Oklahoma
  - University of Texas Southwestern, Dallas, Texas
  - Southwest Rheumatology, Mesquite, Texas
  - University of Utah Health Science center, Salt Lake City, Utah
- Argentina (3):
  - Organizacion Medica de Investigacion, Buenos Aires
  - DOM Centro de Reumatología, Buenos Aires
  - Sanatorio Allende, Córdoba
- Brazil (5):
  - Ser Servicos Especializados Em Reumatologia, Salvador, Estado de Bahia
  - Instituto Pro-Renal, Curitiba, Paraná
  - Hospital das Clinicas - FMUSP Ribeirao Preto, Ribeirão Preto, São Paulo
  - Centro Multidisciplinar de Estudos Clínicos - CEMEC*X*, Santo André, São Paulo
  - Hospital das Clinicas - FMUSP, São Paulo, São Paulo
- Colombia (3):
  - Clinica De La Costa, Barranquilla
  - Hospital Universitario San Ignacio, Bogotá
  - Hospital Pablo Tobon Uribe, Medellín
- France (5):
  - Hopital Henri Mondor, Créteil
  - Hopital Claude Huriez, Lille
  - Groupe Hospitalier Pitie-Salpetriere, Paris
  - Hopital Bichat Claude Bernard, Paris
  - Hopital Rangueil, Toulouse
- Germany (6):
  - Charité Campus Mitte, Med.Klinik, Rheumatologie und Klinische Immunologie, Berlin
  - Städtisches Klinik Dresden-Friedrichstadt, Dresden
  - Universitätsklinikum "Carl Gustav Carus", Dresden
  - Universitätsklinikum Freiburg, Freiburg im Breisgau
  - Universitaetsmedizin Johannes Gutenberg, Mainz
  - Universitätskrankenhaus Tübingen, Tübingen
- Israel (4):
  - Meir Medical Center, Kfar Saba
  - Rabin MC- Belinson campus, Petah Tikva
  - Chaim Sheba Medical Center, Ramat Gan
  - Sourasky Medical Centre, Tel Aviv
- Italy (5):
  - Policlinico di Bari, Bari, Apulia
  - Ospedale Policlinico San Martino, Genoa, Liguria
  - A.O. Spedali Civili Di Brescia-P.O. Spedali Civili, Brescia, Lombardy
  - Azienda Ospedaliera Universitaria Careggi, Florence, Tuscany
  - Azienda Ospedaliera di Padova, Padua, Veneto
- Mexico (3):
  - Centro de Investigación y Tratamiento Reumatológico S.C., Mexico City, Mexico CITY (federal District)
  - Instituto Nacional de Ciencias Médicas Y de La Nutricion Zubirán, Mexico City, Mexico CITY (federal District)
  - Hospital Universitario, Monterrey, Nuevo León
- Peru (5):
  - Instituto Peruano del Hueso y la Articulación, Lima
  - Clínica San Juan Bautista CSJB, Lima
  - Instituto del Cerebro y la Columna Vertebral SAC, Lima
  - Instituto de Ginecología y Reproducción, Lima
  - Hospital Nacional Cayetano Heredia, San Martín de Porres
- Poland (7):
  - Uniwersytecki Szpital Kliniczny nr 4 w Lublinie, Lublin
  - Medyczne Centrum Hetmanska, Poznan
  - Ortopedyczno Rehab Szpital Klinic im Wiktora Degi UM, Poznan
  - Szpital Kliniczny Dzieciatka Jezus, Warsaw
  - Rheuma Medicus Zaklad Opieki Zdrowotnej, Warsaw
  - Narodowy Instytut Geriatrii, Reumatologii i Rehabilitacji im. Prof. Eleonory Reicher, Warsaw
  - Uniwersytecki Szpital Kliniczny im. Jana Mikulicza-Radeckiego we Wroclawiu, Wroclaw
- Russia (4):
  - Federal State Budgetary Scientific Institution Research Institute of Rheumatology V.A. Nasonova, Moscow, Moscow Oblast
  - Federal Centre of Heart, Blood and Endocrinology n.a. V.A.Almazov, Saint Petersburg, Sankt-Peterburg
  - ?Kazan (Privolzhsky) Federal University?, Kazan', Tatarstan Republic
  - SBEI HPE "The First St.Petersburg State Medical University n.a. acad. I.P.Pavlova"of MoH of RF, Saint Petersburg
- Groote Schuur Hospital and University of Cape Town, Cape Town, South Africa
- Spain (4):
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Clinic i Provincial, Barcelona
  - Hospital Ramon y Cajal, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
- Cambridge University Hospitals NHS Foundation Trust - Addenbrookes Hospital, Cambridge, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing

REFERENCES:
- [Derived] Furie RA, Rovin BH, Garg JP, Santiago MB, Aroca-Martinez G, Zuta Santillan AE, Alvarez D, Navarro Sandoval C, Lila AM, Tumlin JA, Saxena A, Irazoque Palazuelos F, Raghu H, Yoo B, Hassan I, Martins E, Sehgal H, Kirchner P, Ross Terres J, Omachi TA, Schindler T, Pendergraft WF 3rd, Malvar A; REGENCY Trial Investigators. Efficacy and Safety of Obinutuzumab in Active Lupus Nephritis. N Engl J Med. 2025 Apr 17;392(15):1471-1483. doi: 10.1056/NEJMoa2410965. Epub 2025 Feb 7. PMID 39927615
- [Derived] Avasare R, Drexler Y, Caster DJ, Mitrofanova A, Jefferson JA. Management of Lupus Nephritis: New Treatments and Updated Guidelines. Kidney360. 2023 Oct 1;4(10):1503-1511. doi: 10.34067/KID.0000000000000230. PMID 37528520
- [Derived] Dossier C, Hogan J. Response to Majeranowski. Pediatr Nephrol. 2021 Jun;36(6):1653. doi: 10.1007/s00467-021-04982-4. Epub 2021 Mar 10. No abstract available. PMID 33693991

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 271 participants with International Society of Nephrology/ Renal Pathology Society (ISN/RPS) 2003 Class III or IV lupus nephritis (LN) treated with standard-of-care (SOC) therapy took part in the study across 72 sites in 15 countries.
  This study consists of blinded treatment with obinutuzumab or placebo, followed by open-label treatment (OLT) with obinutuzumab.
Pre-assignment Details: Participants were randomized in a 1:1 ratio to Obinutuzumab/placebo. As pre-specified in the statistical analysis plan (SAP), participant flow data for all participants randomized to 1 of the 2 dosing schedules of obinutuzumab (Groups 1 & 2) were reported in the combined obinutuzumab treatment group. This study is ongoing.
Groups:
- Obinutuzumab: Participants received obinutuzumab, 1000 milligrams (mg) as an intravenous (IV) infusion on Day 1 and Weeks 2, 24, 26, and either Weeks 50 and 52 or Week 52 only, along with mycophenolate mofetil (MMF) and SOC therapy. Placebo was administered at Week 50 for participants not treated with obinutuzumab. Participants with adequate response at Week 76 continued to receive obinutuzumab at Week 80 and every 6 months (Q6M) thereafter. The dose of MMF can be adjusted at the investigator's discretion beginning at Week 80.
- Placebo: Participants received Obinutuzumab matching placebo as an IV infusion on Day 1 and Weeks 2, 24, 26, 50, and 52. Participants also received SOC therapy and MMF. Participants with adequate response at Week 76 continued to receive placebo at Week 80 and Q6M thereafter. The dose of MMF can be adjusted at the investigator's discretion beginning at Week 80.
Period: Overall Study
Arm/Group | Obinutuzumab | Placebo
Started | 135 | 136
Safety Population (Safety evaluable population included all participants who received any part of blinded infusion of Obinutuzumab/placebo & are grouped according to treatment they received. 3 participants from placebo arm were excluded from the safety analysis as they received no treatment post-randomization. 1 participant randomized to the placebo arm received obinutuzumab & was included in the obinutuzumab arm for safety analysis.) | 136 | 132
Completed Week 76 Assessment | 122 | 120
Completed | 0 | 0
Not Completed | 135 | 136
Not completed — Adverse Event | 1 | 1
Not completed — Death | 5 | 4
Not completed — Lack of Efficacy | 1 | 2
Not completed — Lost to Follow-up | 1 | 2
Not completed — Non-compliance with Study Drug | 1 | 0
Not completed — Reason not Specified | 0 | 5
Not completed — Physician Decision | 0 | 6
Not completed — Withdrawal by Subject | 10 | 14
Not completed — Ongoing in the Study | 116 | 102

BASELINE CHARACTERISTICS:
Population: Efficacy population included all randomized participants regardless of whether they received study drug. As pre-specified in the SAP, demographic and baseline characteristics were to be provided for obinutuzumab (combined treatment groups) and placebo groups.
Groups:
- Obinutuzumab: Participants received obinutuzumab, 1000 mg as an IV infusion on Day 1 and Weeks 2, 24, 26, and either Weeks 50 and 52 or Week 52 only, along with MMF and SOC therapy. Placebo was administered at Week 50 for participants not treated with obinutuzumab. Participants with adequate response at Week 76 continued to receive obinutuzumab at Week 80 and Q6M thereafter. The dose of MMF can be adjusted at the investigator's discretion beginning at Week 80.
- Placebo: Participants received Obinutuzumab matching placebo as an IV infusion on Day 1 and Weeks 2, 24, 26, 50, and 52. Participants also received SOC therapy and MMF. Participants with adequate response at Week 76 continued to receive placebo at Week 80 and Q6M thereafter.
- Total: Total of all reporting groups
Arm/Group | Obinutuzumab | Placebo | Total
Number analyzed (Participants) | 135 | 136 | 271
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.0 (10.5) | 32.7 (10.0) | 32.9 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 114 | 115 | 229
  Male | 21 | 21 | 42
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 71 | 85 | 156
  Not Hispanic or Latino | 54 | 48 | 102
  Unknown or Not Reported | 10 | 3 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 25 | 26 | 51
  Asian | 9 | 7 | 16
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 20 | 20 | 40
  White | 65 | 64 | 129
  More than one race | 11 | 9 | 20
  Unknown or Not Reported | 5 | 10 | 15

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Complete Renal Response (CRR)
Description: CRR was defined as an achievement of all the following criteria: urinary protein-to-creatinine ratio (UPCR) <0.5 gram/gram (g/g); estimated glomerular filtration rate (eGFR) >=85% of baseline, as calculated using the chronic kidney disease epidemiology collaboration (CKD-EPI) equation and no occurrence of intercurrent events of rescue therapy, treatment failure, death or early study withdrawal. Obinutuzumab and placebo were compared using Cochran-Mantel-Haenszel (CMH) test adjusting for the stratification factors region and race. Missing data was imputed by multiple imputations using fully conditional specification (FCS) predicted mean matching method. Percentage have been rounded off.
Time Frame: At Week 76
Population: Efficacy population included all randomized participants regardless of whether they received study drug. As pre-specified in the SAP, all the endpoints were to be compared between the obinutuzumab (combined treatment groups) and placebo groups.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Obinutuzumab | Placebo
Number analyzed (Participants) | 135 | 136
percentage of participants | 46.4 [37.95 to 54.86] | 33.1 [25.18 to 41.00]
Statistical Analysis 1: Comparison: Obinutuzumab vs Placebo; Test type: Superiority; p = 0.0232, Cochran-Mantel-Haenszel — Test 1 of 7 maintaining a fixed sequence testing for type I error control at two-sided alpha 0.05; Adjusted Difference = 13.40, 95% CI 2-sided [1.95 to 24.84]

2. Secondary Outcome: Percentage of Participants Who Achieve CRR With Successful Prednisone Taper at Week 76
Description: CRR with successful prednisone was defined as the achievement of CRR at Week 76 with no receipt of prednisone >7.5 milligrams per day (mg/day) (or equivalent) from Week 64 through Week 76. CRR was defined as achievement of all the following criteria: UPCR <0.5 g/g; eGFR >=85% of baseline, as calculated using the CKD-EPI equation and no occurrence of intercurrent events of rescue therapy, treatment failure, death or early study withdrawal. Analysis was performed using CMH test adjusting for the stratification factors region and race. Missing data was imputed by multiple imputations using FCS predicted mean matching method. Percentage have been rounded off.
Time Frame: At Week 76
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Obinutuzumab | Placebo
Number analyzed (Participants) | 135 | 136
percentage of participants | 42.7 [34.32 to 51.09] | 30.9 [23.12 to 38.65]
Statistical Analysis 1: Comparison: Obinutuzumab vs Placebo; Test type: Superiority; p = 0.0421, Cochran-Mantel-Haenszel — Test 2 of 7 maintaining a fixed sequence testing for type I error control at two-sided alpha 0.05; Adjusted Difference = 11.88, 95% CI 2-sided [0.57 to 23.18]

3. Secondary Outcome: Percentage of Participants Who Achieve a Proteinuric Response
Description: Proteinuric response was defined as an achievement of all the following criteria: UPCR <0.8 g/g and no occurrence of intercurrent events of rescue therapy, treatment failure, death or early study withdrawal. Analysis was performed using CMH test adjusting for the stratification factors region and race. Missing data was imputed by multiple imputations using FCS predicted mean matching method. Percentage have been rounded off.
Time Frame: At Week 76
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Obinutuzumab | Placebo
Number analyzed (Participants) | 135 | 136
percentage of participants | 55.5 [47.09 to 63.95] | 41.9 [33.62 to 50.20]
Statistical Analysis 1: Comparison: Obinutuzumab vs Placebo; Test type: Superiority; p = 0.0227, Cochran-Mantel-Haenszel — Test 3 of 7 maintaining a fixed sequence testing for type I error control at two-sided alpha 0.04 with fallback method; Adjusted Difference = 13.68, 95% CI 2-sided [2.01 to 25.36]

4. Secondary Outcome: Mean Change in eGFR
Description: Change in eGFR from baseline to Week 76 was analyzed using Analysis of Covariance (ANCOVA) model with covariates baseline eGFR and the stratification factors race and region. Death was considered as an intercurrent event which was handled under composite strategy by imputing data after death with 0. Missing data was imputed by multiple imputations using FCS predicted mean matching method. mL/min/1.73 m^2 = milliliters per minute per 1.73 square meters. Adjusted mean has been reported.
Time Frame: At Week 76
Population: as for outcome 1
Measure: Mean (Standard Error); unit: mL/min/1.73 m^2
Arm/Group | Obinutuzumab | Placebo
Number analyzed (Participants) | 135 | 136
mL/min/1.73 m^2 | 2.31 (2.713) | -1.54 (2.706)
Statistical Analysis 1: Comparison: Obinutuzumab vs Placebo; Test type: Superiority; p = 0.1842, ANCOVA — Test 4 of 7 maintaining a fixed sequence testing for type I error control at two-sided alpha 0.05; Difference in Adjusted Means = 3.84, 95% CI 2-sided [-1.83 to 9.51]

5. Secondary Outcome: Percentage of Participants Who Experience Death or Renal-related Events
Description: Percentage of participants with death or renal-related events were defined as participants with one or more of the following events: Death; Treatment failure; Worsening proteinuria, defined as a confirmed ≥50% increase in UPCR to a value ≥3 g/g; Worsening eGFR, defined as a confirmed ≥30% decrease in eGFR to a value <60. Early study withdrawal due to lack of efficacy was an intercurrent event. Participants experiencing the intercurrent event were considered as participants with events under composite strategy. Analysis was performed using CMH test adjusting for the stratification factors region and race. Missing data was imputed by multiple imputations using FCS predicted mean matching method. Percentages have been rounded off.
Time Frame: From Day 1 to Week 76
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Obinutuzumab | Placebo
Number analyzed (Participants) | 135 | 136
percentage of participants | 18.9 [12.11 to 25.61] | 35.6 [27.50 to 43.78]
Statistical Analysis 1: Comparison: Obinutuzumab vs Placebo; Test type: Superiority; p = 0.0026, Cochran-Mantel-Haenszel — Ranked 5 of 7 in the fixed sequence for type I error control. P-value is nominal as the hierarchical testing stops at the first non-significant endpoint; Adjusted Difference = -16.83, 95% CI 2-sided [-27.42 to -6.23]

6. Secondary Outcome: Percentage of Participants Who Achieve an Overall Renal Response (ORR)
Description: ORR was defined as achievement of either CRR or PRR. CRR was defined as achievement of all of the criteria: UPCR <0.5 g/g; eGFR ≥85% of baseline, as calculated using the CKD-EPI equation. PRR was defined as achievement of all of the following criteria: ≥50% reduction in UPCR from baseline; UPCR <1 g/g (or <3 g/g if the baseline UPCR was ≥3 g/g); eGFR ≥85% of baseline, as calculated using the CKD-EPI equation and no occurrence of intercurrent events of rescue therapy, treatment failure, death or early study withdrawal. Analysis was performed using CMH test adjusting for the stratification factors region and race. Missing data was imputed by multiple imputations using FCS predicted mean matching method. Percentage have been rounded off.
Time Frame: At Week 50
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Obinutuzumab | Placebo
Number analyzed (Participants) | 135 | 136
percentage of participants | 59.1 [50.80 to 67.43] | 50.7 [42.16 to 59.22]
Statistical Analysis 1: Comparison: Obinutuzumab vs Placebo; Test type: Superiority; p = 0.1670, Cochran-Mantel-Haenszel — Ranked 6 of 7 in the fixed sequence for type I error control; Adjusted Difference = 8.36, 95% CI 2-sided [-3.41 to 20.12]

7. Secondary Outcome: Change From Baseline in Fatigue Assessed Using Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F) Scale
Description: The FACIT-F is a 13-item questionnaire that assesses self-reported fatigue and its impact upon daily activities and function. Participants scored each item on a 5-point scale: 0 (Not at all) to 4 (Very much). The sum of all responses resulted in the FACIT-F score of 0 (worse score) to 52 (better score). Higher scores indicate less fatigue. Change in FACIT-F score from baseline at Week 76 was analyzed using ANCOVA model with covariates baseline FACIT-F score and the stratification factors race and region. Death was considered as an intercurrent event which was handled under composite strategy by imputing FACIT-F score after death with 0. Missing data was imputed by multiple imputations using FCS predicted mean matching method. Adjusted mean has been reported.
Time Frame: At Week 76
Population: as for outcome 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Obinutuzumab | Placebo
Number analyzed (Participants) | 135 | 136
score on a scale | 1.76 (1.223) | 3.11 (1.212)
Statistical Analysis 1: Comparison: Obinutuzumab vs Placebo; Test type: Superiority; p = 0.2991, ANCOVA — Ranked 7 of 7 in the fixed sequence for type I error control; Difference in Adjusted Means = -1.35, 95% CI 2-sided [-3.89 to 1.20]

8. Secondary Outcome: Change in Log-transformed Anti-double-stranded Deoxyribonucleic Acid (Anti-dsDNA) Titer
Description: Anti-dsDNA are types of autoantibodies produced by the immune system and are indicators of lupus. Anti-dsDNA data was log-transformed before analysis. Missing data was imputed by multiple imputations using FCS predicted mean matching method. Analysis was performed using ANCOVA. Death was considered as an intercurrent event which was handled under composite strategy by imputing data after death with upper limit of quantification (ULOQ, 890 international units/milliliter [IU/mL]). Adjusted mean has been reported.
Time Frame: At Week 50
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Log (IU/mL)
Arm/Group | Obinutuzumab | Placebo
Number analyzed (Participants) | 135 | 136
Log (IU/mL) | -0.38 (0.100) | -0.01 (0.099)
Statistical Analysis 1: Comparison: Obinutuzumab vs Placebo; Test type: Superiority; p = 0.0006, ANCOVA — Not type I error controlled; Difference in Adjusted Means = -0.36, 95% CI 2-sided [-0.57 to -0.16]

9. Secondary Outcome: Change in Complement C3
Description: C3 is a marker of inflammation. Analysis was performed using ANCOVA. Death was considered as an intercurrent event which was handled under composite strategy by imputing data after death with lower limit of quantification (LLOQ)/2 under composite strategy. LLOQ at the central lab was set for C3 at 0.100 grams/liters (g/L). Missing data was imputed by multiple imputations using FCS predicted mean matching method. Adjusted mean has been reported.
Time Frame: At Week 50
Population: as for outcome 1
Measure: Mean (Standard Error); unit: g/L
Arm/Group | Obinutuzumab | Placebo
Number analyzed (Participants) | 135 | 136
g/L | 0.20 (0.030) | 0.06 (0.030)
Statistical Analysis 1: Comparison: Obinutuzumab vs Placebo; Test type: Superiority; p < 0.0001, ANCOVA — Not type I error controlled; Difference in Adjusted Means = 0.14, 95% CI 2-sided [0.08 to 0.20]

10. Secondary Outcome: Change in Systematic Lupus Erythematosus Disease Activity Index 2000 (SLEDAI-2K)
Description: The SLEDAI-2K is a 24-item instrument that evaluates clinical symptoms and laboratory markers across nine organ systems and was used to capture changes in lupus-related disease activity. SLE manifestations are assessed by the clinician if present within the last 30 days and added to determine the total SLEDAI-2K score, which ranges from 0 to 105. Higher scores indicate increased disease activity. The analysis was performed using ANCOVA. Death was considered as an intercurrent event which was handled under composite strategy by imputing data after death with 105, the highest possible score. Missing data was imputed by multiple imputations using FCS predicted mean matching method. Adjusted mean has been reported.
Time Frame: At Week 76
Population: as for outcome 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Obinutuzumab | Placebo
Number analyzed (Participants) | 135 | 136
score on a scale | -5.63 (1.456) | -5.51 (1.432)
Statistical Analysis 1: Comparison: Obinutuzumab vs Placebo; Test type: Superiority; p = 0.9384, ANCOVA — Not type I error controlled; Difference in Adjusted Means = -0.12, 95% CI 2-sided [-3.11 to 2.87]

11. Secondary Outcome: Time to Onset of CRR
Description: CRR was defined as an achievement of all the following criteria: UPCR <0.5 g/g; eGFR >=85% of baseline, as calculated using the CKD-EPI equation and no occurrence of intercurrent events of rescue therapy, treatment failure, death or early study withdrawal. Participants who experienced the intercurrent events before achieving CRR as well as participants who completed 76-week treatment period without experiencing CRR were censored at Week 76. Summary statistics of time to onset of CRR are Kaplan-Meier estimates. A log-rank test was used to compare obinutuzumab and placebo. The median time to onset of CRR was greater than Week 76 due to considering the upper limit of the Week 76 analysis visit window in this analysis. The upper limit of the Week 76 visit window was 3 days prior to the next obinutuzumab or placebo infusion or 30 days beyond Week 76 whichever is shorter.
Time Frame: From baseline (Day 1) up to 80.3 weeks
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Obinutuzumab | Placebo
Number analyzed (Participants) | 135 | 136
weeks | 76.4 [76.1 to 77.4] | 80.3 [76.3 to NA] — Upper limit of 95% CI was not estimable due to an insufficient number of participants with events.
Statistical Analysis 1: Comparison: Obinutuzumab vs Placebo; Test type: Superiority; p = 0.1324, Log Rank — Not type I error controlled; Hazard Ratio (HR) = 1.31, 95% CI 2-sided [0.91 to 1.89]

12. Secondary Outcome: Percentage of Participants Who Achieve CRR With Serum Creatinine Criteria
Description: CRR with serum creatinine criteria was defined as achievement of all the following criteria: UPCR <0.5 g/g; Serum creatinine ≤ ULN, as determined by the central laboratory; serum creatinine not increased from baseline by > 25% and no occurrence of intercurrent events of rescue therapy, treatment failure, death or early study withdrawal. Analysis was performed using CMH test adjusting for the stratification factors region and race. Percentage have been rounded off.
Time Frame: At Week 76
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Obinutuzumab | Placebo
Number analyzed (Participants) | 135 | 136
percentage of participants | 46.4 [37.90 to 54.85] | 33.1 [25.18 to 41.00]
Statistical Analysis 1: Comparison: Obinutuzumab vs Placebo; Test type: Superiority; p = 0.0237, Cochran-Mantel-Haenszel — Not type I error controlled; Adjusted Difference = 13.37, 95% CI 2-sided [1.91 to 24.82]

13. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: An AE was any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An AE can therefore be any unfavorable and unintended sign (including abnormal laboratory values or abnormal clinical test results), symptoms, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product.
Time Frame: Up to Week 76
Population: Safety evaluable population included all participants who received any part of blinded infusion of obinutuzumab or placebo and were grouped according to the treatment they actually received rather than the treatment assigned. As pre-specified in the SAP, safety data were to be provided for obinutuzumab (combined treatment groups) and placebo groups.
Measure: Count of Participants; unit: Participants
Arm/Group | Obinutuzumab | Placebo
Number analyzed (Participants) | 136 | 132
Participants | 126 | 117

14. Secondary Outcome: Number of Participants With Adverse Events of Special Interest (AESIs)
Description: An AE was any untoward medical occurrence in participant administered a pharmaceutical product & which does not necessarily have to have a causal relationship with treatment. It can therefore be any unfavorable & unintended sign (including abnormal laboratory values/ abnormal clinical test results), symptoms, or disease temporally associated with use of pharmaceutical product, whether or not considered related to product. AESIs included potential drug-induced liver injury that include an elevated alanine transaminase (ALT) & aspartate aminotransferase (AST) in combination with either an elevated bilirubin or clinical jaundice defined by Hy's law; suspected transmission of an infectious agent by study drug; infusion-related reactions (IRRs); grade 3/higher infections; any hepatitis B reactivation and progressive multifocal leukoencephalopathy (PML); drug-related neutropenia; drug-related thrombocytopenia; gastrointestinal perforations and worsening of pre-existing cardiac conditions
Time Frame: Up to Week 76
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Obinutuzumab | Placebo
Number analyzed (Participants) | 136 | 132
Participants
  IRRs | 21 | 15
  Grade 3-5 infection | 21 | 9
  Any Hepatitis B reactivation and PML | 0 | 0
  Drug related Neutropenia | 17 | 5
  Drug related Thrombocytopenia | 1 | 0
  Gastrointestinal Perforations | 0 | 0
  Worsening of pre-existing Cardiac Conditions | 0 | 2
  Hy's Law | 0 | 0
  Suspected Transmission of an Infectious Agent by the Study Drug | 0 | 0

15. Secondary Outcome: Number of Participants With Anti-Drug Antibodies (ADAs) Positive Post-Treatment
Description: Determination of anti-obinutuzumab antibodies in serum samples were performed using a validated enzyme-linked Immunosorbent Assay (ELISA) method. Participants were considered to be ADA positive if they were ADA negative or have missing data at baseline but develop an ADA response following study drug exposure (treatment-induced ADA response), or if they were ADA positive at baseline and the titer of one or more post baseline samples was at least ≥ 4-fold greater than the titer of the baseline sample (treatment-enhanced ADA response).
Time Frame: Up to approximately 11 years
Reporting Status: Not Posted, anticipated posting 2029-02

16. Secondary Outcome: Total Peripheral B-Cell (CD19) Count
Time Frame: Up to approximately 11 years
Reporting Status: Not Posted, anticipated posting 2032-02

17. Secondary Outcome: Concentration of Obinutuzumab in Serum
Time Frame: Up to approximately 11 years
Reporting Status: Not Posted, anticipated posting 2032-02

ADVERSE EVENTS:
Time Frame: Up to Week 76 Data collected up to the primary completion date (Up to Week 76) is reported. Data collection post Week 76 is still ongoing. Final data will be reported 1 year after the study completion date. As pre-specified in the SAP, safety data were to be provided for obinutuzumab (combined treatment groups) and placebo groups. AE data were collected for all Obinutuzumab participants together, without regard to or information of the specific Obinutuzumab group participants they were part of.
Description: Safety evaluable population=all participants who received any part of blinded infusion of Obinutuzumab/placebo & are grouped according to treatment they received. 3 participants from placebo arm did not receive treatment & were excluded from the safety analysis. 1 participant randomized to placebo arm received obinutuzumab & was included in obinutuzumab arm for safety analysis. Includes AEs until point of rescue for participants who received rescue therapy (except corticosteroid-only rescue).
Arm/Group | Obinutuzumab | Placebo
All-Cause Mortality (participants affected / at risk) | 5/136 | 4/132
Serious Adverse Events (participants affected / at risk) | 44/136 | 24/132
Other Adverse Events (participants affected / at risk) | 107/136 | 94/132
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Obinutuzumab (N=136) | Placebo (N=132)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 4 (7) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1)
Scintillating scotoma (Eye disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Anal inflammation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis erosive (Gastrointestinal disorders) | 0 (0) | 1 (1)
Large intestinal stenosis (Gastrointestinal disorders) | 1 (2) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (2) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 2 (2)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Bacterial diarrhoea (Infections and infestations) | 0 (0) | 1 (1)
Bacterial infection (Infections and infestations) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 4 (4) | 1 (1)
COVID-19 pneumonia (Infections and infestations) | 7 (8) | 0 (0)
Device related bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 3 (3) | 2 (2)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 1 (1)
Peritonsillar abscess (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 4 (4) | 3 (3)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 0 (0)
Post-acute COVID-19 syndrome (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Tooth abscess (Infections and infestations) | 1 (1) | 0 (0)
Urethritis (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 4 (4) | 2 (2)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0)
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 1 (1) | 0 (0)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Vulvovaginal warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Autoimmune encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 3 (4) | 2 (2)
Nephrotic syndrome (Renal and urinary disorders) | 1 (1) | 2 (2)
Proteinuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Cervical dysplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Hypertensive urgency (Vascular disorders) | 0 (0) | 1 (1)
Peripheral venous disease (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Obinutuzumab (N=136) | Placebo (N=132)
Anaemia (Blood and lymphatic system disorders) | 7 (7) | 9 (10)
Leukopenia (Blood and lymphatic system disorders) | 7 (10) | 6 (8)
Neutropenia (Blood and lymphatic system disorders) | 12 (14) | 4 (5)
Abdominal pain (Gastrointestinal disorders) | 4 (6) | 10 (16)
Diarrhoea (Gastrointestinal disorders) | 28 (33) | 21 (35)
Nausea (Gastrointestinal disorders) | 8 (9) | 11 (15)
Vomiting (Gastrointestinal disorders) | 10 (14) | 11 (12)
Pyrexia (General disorders) | 4 (5) | 8 (8)
Bronchitis (Infections and infestations) | 13 (13) | 11 (12)
COVID-19 (Infections and infestations) | 35 (40) | 30 (32)
Gastroenteritis (Infections and infestations) | 5 (7) | 10 (14)
Herpes zoster (Infections and infestations) | 9 (11) | 7 (7)
Influenza (Infections and infestations) | 6 (7) | 7 (7)
Nasopharyngitis (Infections and infestations) | 10 (13) | 9 (11)
Upper respiratory tract infection (Infections and infestations) | 16 (22) | 13 (24)
Urinary tract infection (Infections and infestations) | 19 (27) | 15 (20)
Infusion related reaction (Injury, poisoning and procedural complications) | 19 (22) | 14 (18)
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 (9) | 10 (11)
Back pain (Musculoskeletal and connective tissue disorders) | 7 (7) | 5 (5)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 (3) | 7 (7)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3) | 7 (7)
Headache (Nervous system disorders) | 12 (13) | 8 (12)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (8) | 2 (2)
Hypertension (Vascular disorders) | 8 (8) | 9 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2024-02-07): https://cdn.clinicaltrials.gov/large-docs/77/NCT04221477/Prot_000.pdf
  • Statistical Analysis Plan (2024-07-19): https://cdn.clinicaltrials.gov/large-docs/77/NCT04221477/SAP_001.pdf